CLINICAL TRIAL: NCT00771511
Title: Cervical Capsaicin for Labor Induction and Pain Relief
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never started
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Pamela Flood, Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAD5899
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Labor Pain; Pregnancy Loss; Labor Induction
MeSH Terms: conditions — Labor Pain | interventions — Capsaicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Capsaicin cream applied to cervix after lidocaine gel
  Interventions: Drug: capsaicin
- 2 (Placebo Comparator): only lidocaine applied to the cervix
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: capsaicin — capsaicin cream 0.1% 10 ml applied to cervix
  Arms: 1
Drug: Placebo — Only lidocaine gel will be appled to the cervix
  Arms: 2

SUMMARY:
In the setting of fetal demise it is important to help the mother deliver the fetus expeditiously and with as little physical trauma as possible. This study hypothesizes that application of capsaicin to the uterine cervix will enhance cervical ripening and desensitize pain fibers such that delivery is less painful.

DETAILED DESCRIPTION:
Induction of labor is associated with increased risk of cesarean section and elevated pain when compared to labor of spontaneous onset. In the setting of intrauterine fetal demise (IUFD), it is desirable to induce labor in order to achieve a successful vaginal delivery for the health and well being of the mother, thereby avoiding operative fetal extraction.

The current protocol for midtrimester labor induction prior to 24 weeks gestational age includes intravaginal cytotec(misoprostol) 200 mcg every 6 hours for up to 24 hours, occasionally followed by oxytocin infusion. When an IUFD occurs at 24 or greater weeks gestational age, labor is induced with cytotec 25 or 50 mcg every 4 hours and/or oxytocin infusion. The investigators hypothesize that application of lidocaine to the uterine cervix followed by 0.1% capsaicin cream will facilitate cervical ripening and decrease the pain of labor induction when compared to use of a placebo cream. Capsaicin 8methylNvannilyl6nonenamide) activates TRPV1, a nonselective cation channel activated directly by heat, and low pH, and indirectly by a number of inflammatory factors, including nerve growth factor (NGF), bradykinin, lipids, and prostaglandins. Activation of TRPV1 by capsaicin results in an influx of Ca2 and Na ions, depolarization, exocytosis of neuropeptides and excitatory amino acids, and induces a burning sensation. This initial phase is followed by prolonged desensitiztion that is dose dependent. Once the TRPV1 receptor is desensitized, pain transmission through Ctype primary afferent receptors is reduced. The pain relief from capsaicin is due to desensitization of the TRPV1 receptor. The enhancement of cervical ripening is due to activation of primary afferent Cfibers, release of neuropeptides substance P, neurokinin A, calcitonin generelated peptide, secretoneurin and nitric oxide to help orchestrate a series of local inflammatory responses including vasodilation, vascular permeability with tissue edema and protein extravasation, and migration of inflammatory immune cells. In a study of pregnant rats, vaginal lidocaine gel was applied followed by capsaicin sham cream. A blinded observer monitored behavior via video over the next 72 hours. All animals treated with capsaicin delivered on day 22 with minimal pain behaviors while 90% of sham treated animals delivered as expected on day 23 with normal pain related behavior. All pups were delivered live and rearing and suckling behavior was normal.

ELIGIBILITY:
Inclusion Criteria:

* IUFD after 20 weeks gestation

Exclusion Criteria:

* Chorioamnionitis
* Chronic pain syndrome
* Current pain meds during pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10 (Estimated); Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Pain report during labor | 48 hours after labor induction

SECONDARY OUTCOMES:
Bishop's score | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Flood, MD, Principal Investigator — Columbia University